CLINICAL TRIAL: NCT00200616
Title: Antimicrobial Prophylaxis in Children With Isolated Vesico-Ureteral Reflux. A Randomised Prospective Study of Continuous Low Dose of Trimethoprim-Sulfamethoxazole Versus Surveillance.
Brief Title: Usefulness of Antimicrobial Prophylaxis in Children With Isolated Vesico-Ureteral Reflux.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Claude GUYOT, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/00/10-O
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Urinary Tract Infection
Keywords: Urinary tract infection; Vesico-renal reflux; Child; Antimicrobial prophylaxis; Recurrence of urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Antimicrobial prophylaxis

SUMMARY:
Randomized, prospective, multicenter study in order to assess the usefulness of antimicrobial prophylaxis in children with isolated vesico-ureteral reflux (grade III or less).

DETAILED DESCRIPTION:
A voiding cystourethrogram was performed for each child less than 3 years old with a first urinary tract infection. In case of vesico-ureteral reflux, a randomization was done between continuous antimicrobial prophylaxis with low dose of trimethoprim-sulfamethoxazole and no antibioprophylaxis. Duration of follow up was 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 3 years old
* First proved urinary tract infectionIsolated vesico-ureteral reflux
* Parents have been fully informed and have given written informed consent to participate in the study

Exclusion Criteria:

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232
Dates: Start 2001-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
End point : recurrence of urinary tract infection during the study period (0 è 18 months)

SECONDARY OUTCOMES:
1) Type of urinary tract infection (pyelonephritis or cystitis)
2) Evaluation of the quality of life with a validated questionnaire done at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Claude GUYOT, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France